CLINICAL TRIAL: NCT03137485
Title: Management of Lumbar Postero-lateral Single Level Disc Herniation: Comparative Study Between Conventional and Endoscopic Lumbar Discectomy
Brief Title: Comparison Between Conventional vs. Endoscopic Lumbar Discectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, H A Othman, Resident Doctor, Neurosurgery Department, Assiut Universiy Hosipitals, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDODISC
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Lumbar Disc Herniation
Keywords: lumbar disc herniation; endoscopic discectomy; open discectomy; comparative study; Translaminar; surgery
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Patients in this arm will have conventional open lumbar discectomy operation.
  Interventions: Procedure: Conventional open lumbar discectomy
- Endoscopic (Active Comparator): Patients in this arm will have Percutaneous Endoscopic Translaminar lumbar discectomy operation using Easy Go system Endoscopy
  Interventions: Procedure: Percutaneous Endoscopic Translaminar lumbar discectomy.; Device: Easy Go system Endoscopy

INTERVENTIONS:
Procedure: Conventional open lumbar discectomy — Removal of single level lumbar disc herniation through conventional discectomy.
  Arms: Conventional
Procedure: Percutaneous Endoscopic Translaminar lumbar discectomy. — Removal of single level Lumbar disc herniation using endoscope.
  Arms: Endoscopic
Device: Easy Go system Endoscopy — This system will be used to remove herniated disc in endoscopic group
  Arms: Endoscopic

SUMMARY:
This study is aimed to compare between the results of conventional lumbar discectomy and the newly used technique in our department; endoscopic lumbar discectomy in neurosurgery department Assiut university hospitals, so that we can offer our patients the best service in an updated and minimally invasive way.

DETAILED DESCRIPTION:
Lumbar discectomy is one of the most common operation performed worldwide for lumbar-related symptoms. Lumbar disc herniation accounts for only 5% of all low back pain problems but is the most common cause of radiating nerve root pain, sciatica.

Mixter and Barr described the first surgical procedure to remove the herniated lumbar disc in 1934 through a laminectomy and durotomy, with later enhancement by Semmes, who described approaching the herniated disc through hemilaminectomy and retraction of the dural sac. This became popularized as the "classical discectomy technique.

During the latter half of the 19th century, more techniques were developed to remove the herniated disc with minimal invasiveness. The first herniated disc excision using a microscope (microdiscectomy) was performed by Yasargil in 1977, which was the standard surgical procedure at the time In 1993, Mayer and Brock and then in 1997, Smith and Foley described endoscopic discectomy techniques. With these minimally invasive techniques, authors demonstrated decreased soft tissue manipulation, operative time, blood loss, and hospital stay, allowing early recovery.

In this study we try to evaluate clinical and radiological outcomes of percutaneous endoscopic translaminar discectomy at our hospital.

ELIGIBILITY:
Inclusion Criteria:

* single level, postero-lateral, denovo lumbar disc herniation including those with migrated and/or sequestrated discs.
* L4,5 &L5,S1 disc prolapse
* Failure of conservative management after 12 weeks.

Exclusion Criteria:

* central, far lateral, recurrent and/or multiple level disc herniation.
* Lateral recess stenosis or spondylolisthesis.
* presence of neurological deficit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Improvement of Preoperative low back pain and radicular pain. | Up to ten months post operative.
  Improvement of preoperative low back pain and radicular pain.Clinical outcomes will be measured using Visual Analogue Scale.
Functional Improvement | Up to ten months post operative.
  Functional Improvement using modified MacNab's criteria

SECONDARY OUTCOMES:
Hospital stay. | up to one week.
  Time spent in hospital post operative.
Periprocedural complication. | Up to two weeks.
  Such as neurological deficit, Cerebro-Spinal fluid (CSF) leak, wound infection...etc.
Blood loss | intraoperative.
  Amount of blood loss intraoperative.
lumbo-sacral MRI | Up to six months
  Demonstration of any disc herniation recurrence.
Operative time | Intraoperative
  duration of operation
Wound length | Intraoperative
  Length of incision needed by surgeon to complete each approach

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad T Ahmed, Professor, Study Chair — Head of Neurosurgery Department, Assiut University Hospitals

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gibson JN, Waddell G. Surgical interventions for lumbar disc prolapse. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD001350. doi: 10.1002/14651858.CD001350.pub4. PMID 17443505
- [Background] Gotfryd A, Avanzi O. A systematic review of randomised clinical trials using posterior discectomy to treat lumbar disc herniations. Int Orthop. 2009 Feb;33(1):11-7. doi: 10.1007/s00264-008-0559-2. Epub 2008 May 24. PMID 18500517
- [Background] Evaniew N, Khan M, Drew B, Kwok D, Bhandari M, Ghert M. Minimally invasive versus open surgery for cervical and lumbar discectomy: a systematic review and meta-analysis. CMAJ Open. 2014 Oct 1;2(4):E295-305. doi: 10.9778/cmajo.20140048. eCollection 2014 Oct. PMID 25485257
- [Background] Jiang W, Sun B, Sheng Q, Song X, Zheng Y, Wang L. Feasibility and efficacy of percutaneous lateral lumbar discectomy in the treatment of patients with lumbar disc herniation: a preliminary experience. Biomed Res Int. 2015;2015:378612. doi: 10.1155/2015/378612. Epub 2015 Jan 28. PMID 25695066